CLINICAL TRIAL: NCT03552718
Title: QUILT-2.025 NANT Neoepitope Yeast Vaccine (YE-NEO-001): Adjuvant Immunotherapy Using a Personalized Neoepitope Yeast-Based Vaccine To Induce T-Cell Responses In Subjects W/ Previously Treated Cancers.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NantBioScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-2.025
Record Dates: First submitted 2018-05-25; First posted 2018-06-12 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Breast Cancer; Head and Neck Squamous Cell Carcinoma; Melanoma; Non Small Cell Lung Cancer; Pancreatic Cancer; Liver Cancer
Keywords: solid tumors
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: NANT Neoepitope Yeast Vaccine (YE-NEO-001) (Experimental)
  Interventions: Biological: YE-NEO-001

INTERVENTIONS:
Biological: YE-NEO-001 — Personalized recombinant yeast-based vaccine engineered to express multiple neoantigen epitopes (neoepitopes) based on an individual subject's tumor molecular profile.
  Other Names: YE-NEO-001 Injectable Suspension

SUMMARY:
This is a phase 1 study to evaluate the safety, the Recommended Phase 2 Dose (RP2D), and preliminary efficacy of a personalized neoepitope yeast-based vaccine, YE-NEO-001, in subjects who have completed potentially curative therapy for their solid cancer and who would otherwise be entering a period of surveillance for recurrent disease.

DETAILED DESCRIPTION:
This is a phase 1 trial to evaluate the safety, the RP2D, and preliminary efficacy of a personalized neoepitope yeast-based vaccine, YE-NEO-001, in subjects who have completed potentially curative therapy for their type of solid cancer (eg, colorectal cancer, breast cancer, head and neck squamous cell carcinoma, melanoma) and would otherwise be entering a period of surveillance for recurrent disease.

The study will be conducted in two parts: part 1 will involve dose escalation, and part 2 will involve the expansion of the RP2D to further evaluate the safety of YE-NEO-001. In part 2 of the study, dose expansion will occur when the RP2D has been determined. An additional 4 subjects may be enrolled in part 2, for a total of up to 10 subjects at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

Pre-treatment Phase: Tissue Procurement and Development of Vaccine

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically-confirmed cancer amenable to treatment with curative intent as part of SoC. Must be willing to provide a tumor tissue sample (either a tumor biopsy specimen or tissue from resected tumor not used for diagnostic purposes) and a blood sample for tumor molecular profiling.

   * Solid cancers include any of the following surgically resectable cancers: colorectal cancer, head and neck squamous cell carcinoma, non-small cell lung cancer, breast cancer (either hormone receptor positive, HER2-positive or negative, or triple-negative breast cancer), pancreatic cancer, liver cancer, and melanoma. Curative therapy, whether surgery, radiation therapy, or adjuvant chemotherapy, must be completed per National Comprehensive Cancer Network (NCCN) guidelines.
4. Must be willing to agree to initiation of development of personalized YE-NEO-001 vaccine.

Treatment Phase:

1. No evidence of disease (NED) at first assessment post multi-modality therapy (ie, surgery and/or radiation therapy and/or chemotherapy). Subjects treated with definitive radiation therapy are considered NED if they have no evidence of cancer growth on the first and second surveillance CT scans. Subjects who have disease recurrence prior to the start of the vaccination process are also eligible if no satisfactory alternative treatment options are available or if subject has refused all other available therapies.
2. Must have received < 6 months of SoC therapy.
3. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
4. ECOG performance status of 0 to 2.
5. Must be willing to provide blood samples prior to the start of treatment on this study for exploratory analyses.
6. If cancer recurs while on treatment on this study, must be willing to provide a tumor biopsy specimen for exploratory analyses, if considered safe by the Investigator.
7. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
8. Agreement to practice effective contraception for female subjects with child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, IUDs, and abstinence.

Exclusion Criteria:

Pre-treatment Phase: Tissue Procurement and Development of Vaccine

1. Unable or unwilling to attend required study visits and return for adequate follow-up, as required by this protocol.

Treatment Phase:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Active autoimmune disease requiring systemic immunosuppressive treatment within 4 weeks prior to enrollment on this study (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma, ankylosing spondylitis, scleroderma, multiple sclerosis). A history of inactive autoimmune disease or autoimmune disease not requiring systemic immunosuppressive therapy within 4 weeks prior to study enrollment is allowed.
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. ANC < 1,000 cells/mm^3.
   2. Platelet count < 75,000 cells/mm^3.
   3. Uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
   4. Total bilirubin > ULN (unless the subject has documented Gilbert's syndrome).
   5. AST (SGOT) or ALT (SGPT) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or > 10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Positive results of screening test for HIV.
8. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
9. Known hypersensitivity to any component of the study medication(s).
10. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with the study treatment. Anti-androgen and anti-estrogen medications are allowed.
11. Participation in an investigational drug study or history of receiving any investigational treatment within 30 days prior to initiation of treatment on this study, except for testosterone-lowering therapy in men with prostate cancer.
12. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
13. Concurrent participation in any interventional clinical trial.
14. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 19 months
Recommended Phase 2 Dose | 19 months

SECONDARY OUTCOMES:
Recurrence rate | 19 months
  The appearance of any lesion that is confirmed by biopsy (in subjects with no evidence of disease (NED) at the start of the treatment only)
Disease-free survival (DFS) | 24 months
  The time from the date of first YE-NEO-001 treatment to the date of disease recurrence or death (any cause), whichever occurs first (in subjects with NED at the start of treatment only)
Overall survival (OS) | 36 months
  The time from the date of first YE-NEO-001 treatment to the date of death (any cause) (in all subjects)
Progression-free survival (PFS) | 24 months
  The time from the date of first YE-NEO-001 treatment to the date of disease progression or death (any cause), whichever occurs first (in all subjects)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: Undecided